CLINICAL TRIAL: NCT06896942
Title: EVALUATION OF A COMMUNITY DRIVEN, EQUITABLE INTERVENTION FOR BLACK CHILDREN WITH AUTISM
Brief Title: Autism Doula Program Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0473; UL1TR001425 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Health Equity; Autism Spectrum Disorder
Keywords: health equity; autism spectrum disorder; family navigation
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This pilot study will obtain and compare data from the intervention group (i.e., families receiving Autism Doula services) and the control group (i.e., families receiving care as usual including DDBP Family Navigation) to examine the acceptability, feasibility, and preliminary effectiveness of an Autism Doula program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Autism doula care includes providing caregivers with culturally-responsive support, helping them navigating next steps for their child's care, connecting them with the Black autism community, and providing services to alleviate caregiver stress (e.g., cooking, cleaning, respite care).
  Interventions: Other: Autism Doula
- Control group (Active Comparator): The control group will receive care as usual and a referral to DDBP family navigation, which is usually a one time telehealth appointment to plan next steps for their child's care.
  Interventions: Other: DDBP Family Navigation

INTERVENTIONS:
Other: Autism Doula — The Autism Doula provides caregiver support, navigation with next steps for their child, connects families to resources and the Black autism community, and coordinates services to help alleviate caregiver stress (e.g., cleaning, cooking, respite care).
  Arms: Intervention Group
Other: DDBP Family Navigation — A one-time consult with a DDBP family navigator via telehealth to come up with an action plan for next steps for the patient's care.
  Arms: Control group

SUMMARY:
Background: Findings from a group level assessment with caregivers of Black children with autism revealed barriers to equitable care and services (e.g., a lack of cultural representation among their child's care team, caregiver stress, stigma, and uncertainty about services needed). The Autism Doula program was identified by the community to address the aforementioned barriers and provide culturally matched family navigation and social-emotional support while also acknowledging the unique experiences and values of caregivers of Black children with autism.

Impact: The current project aims to assess the acceptability, feasibility, and preliminary effectiveness of the Autism Doula program and promote equitable care for Black children with autism and their families.

Methods: Fifty-six Black families of children 18 months to five years of age who recently received a new diagnosis of autism spectrum disorder from CCHMC will be recruited to the current study. Twenty-six families will be randomly assigned to either the control group (i.e., care as usual including DDBP Family Navigation) or the intervention group (i.e., Autism Doula services). Feasibility and acceptability data will be gathered, including satisfaction of both groups, how many families approached agree to be in the study, how many sessions with the doula were successfully completed, and was the intervention content delivered as intended. Additionally, preliminary effectiveness will be evaluated by examining completion of recommended next steps, caregivers' perceived stress, and self-efficacy.

Implications: Data from this project will provide evidence that the Autism Doula program is feasible, acceptable, and effective, ultimately demonstrating it as an equitable care approach for Black children with autism and their families.

Future Directions: Findings from this pilot project will highlight the need for growth of the Autism Doula program to promote culturally competent care and health equity for Black children with autism and their families.

DETAILED DESCRIPTION:
The current project aims to evaluate a community driven, equitable intervention for Black children with autism. Specifically, we will assess the feasibility and acceptability of the Autism Doula program to enhance culturally responsive care and services for Black children newly diagnosed with autism and their families. The Autism Doula intervention will be measured in several ways, including number of families who complete the Autism Doula intervention, Autism Doula sessions successfully completed, content delivered as intended, and the satisfaction of the families involved in the intervention group. Additionally, preliminary effectiveness will be assessed by comparing the intervention group (i.e., families who receive Autism Doula services) to the experiences of families who receive care as usual including DDBP Family Navigation. Specifically, we will examine caregiver perceived stress levels, caregiver self-efficacy, and initiation of recommended next steps/services. We hypothesize that families receiving Autism Doula services will report high satisfaction with the program and that the program will be determined to be feasible and effective. Should results reveal acceptability, feasibility, and preliminary effectiveness of the Autism Doula intervention, additional funding will be sought out in collaboration with the Division of Developmental and Behavioral Pediatrics (DDBP) at CCHMC to expand the program. Aligned with the hospital wide initiative of incorporating family navigation into clinical care, DDBP leadership has made it a priority to provide culturally-response family navigation, similar to the Autism Doula program.

ELIGIBILITY:
Inclusion Criteria: caregivers of children who are 18 months to five years and recently diagnosed with autism. Caregivers must identify as Black and be over the age of 18 and identify their children as Black.

Ages: 18 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Autism Doula field notes | from enrollment to end of doula program at 3 months
  The Autism Doula will have an electronic field note in REDCap that includes the date of contact with family, contact method, and a checklist of intervention content delivered (e.g., assistance with scheduling therapy, contacting early intervention, providing social support). To ensure confidentiality of participants, this REDCap project will be separate from the REDCap project for study measures.
Satisfaction Survey | end of the autism doula program at 3 months after enrollment
  This survey will be given following completion of the Autism Doula program or at three months for the control group. This survey will have two versions, one for the Autism Doula program and one for DDBP Family Navigation, and was adapted from the Patient Satisfaction with Logistical Aspects of Navigation Scale (PSN-L). Questions will be asked on a Likert Scale from 1 (strongly disagree) to 5 (strongly agree) and include their satisfaction with the services they received from the Autism Doula. The items are summed for a total score and higher scores indicate higher satisfaction. There will also be a comment section for open-ended feedback.
Chart Review Form: | end of the autism doula program at 3 months after enrollment
  The Chart Review form was developed by research staff and will be used to obtain relevant information pertaining to the completion of recommended next steps, including the following: speech therapy, occupational therapy, Applied Behavior Analysis, Early Intervention services, establishing care with a developmental pediatrician, and behavior therapy. This form will be completed by research staff three months after study enrolment for the control group and after completion of the Autism Doula program for the intervention group (i.e., three months).

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | at study enrollment until after autism doula intervention (3 months)
  The PSS measures perceptions of stress according to how uncontrollable, unpredictable, and overloaded participants view their lives. This 14 item self-report test measures stress from ongoing life circumstances, from anticipating future events, and reactions to specific events. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. The manual for the PSS reports findings supporting the reliability and validity of this measure. This survey will be administered at study enrollment and again three months later for the control group and after completion of the Autism Doula program for the intervention group (i.e., three months).
Early Intervention (EI) Parent Self Efficacy Scale | at study enrollment until after autism doula intervention (3 months)
  This scale is a 16-item scale used to assess EI related competence beliefs of parents of children with disabilities. The manual for this scale reports findings supporting the reliability and validity of this measure. This survey will be administered at study enrollment and again six months later for the control group and after completion of the Autism Doula program for the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: De-identified data will be made available to all those who inquire.

REFERENCES:
- [Background] Hoagwood KE, Cavaleri MA, Serene Olin S, Burns BJ, Slaton E, Gruttadaro D, Hughes R. Family support in children's mental health: a review and synthesis. Clin Child Fam Psychol Rev. 2010 Mar;13(1):1-45. doi: 10.1007/s10567-009-0060-5. PMID 20012893
- [Background] Ogunwole SM, Bennett WL, Williams AN, Bower KM. Community-Based Doulas and COVID-19: Addressing Structural and Institutional Barriers to Maternal Health Equity. Perspect Sex Reprod Health. 2020 Dec;52(4):199-204. doi: 10.1363/psrh.12169. Epub 2021 Jan 5. No abstract available. PMID 33399272
- [Background] Castelin S, Okorodudu J, Smith T. Partnering With a Purpose: Promoting Equity and Justice for Black Children With Autism Spectrum Disorder. J Dev Behav Pediatr. 2024 Jul-Aug 01;45(4):e302-e308. doi: 10.1097/DBP.0000000000001276. Epub 2024 Jul 17. PMID 39023854
- [Background] Smith KA, Gehricke JG, Iadarola S, Wolfe A, Kuhlthau KA. Disparities in Service Use Among Children With Autism: A Systematic Review. Pediatrics. 2020 Apr;145(Suppl 1):S35-S46. doi: 10.1542/peds.2019-1895G. PMID 32238530
- [Background] Shaw KA, Bilder DA, McArthur D, Williams AR, Amoakohene E, Bakian AV, Durkin MS, Fitzgerald RT, Furnier SM, Hughes MM, Pas ET, Salinas A, Warren Z, Williams S, Esler A, Grzybowski A, Ladd-Acosta CM, Patrick M, Zahorodny W, Green KK, Hall-Lande J, Lopez M, Mancilla KC, Nguyen RHN, Pierce K, Schwenk YD, Shenouda J, Sidwell K, Vehorn A, DiRienzo M, Gutierrez J, Hallas L, Hudson A, Spivey MH, Pettygrove S, Washington A, Maenner MJ. Early Identification of Autism Spectrum Disorder Among Children Aged 4 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2020. MMWR Surveill Summ. 2023 Mar 24;72(1):1-15. doi: 10.15585/mmwr.ss7201a1. PMID 36952289
- [Background] Fisher AP, Lynch JD, Jacquez FM, Mitchell MJ, Kamimura-Nishimura KI, Wade SL. A systematic review examining caregivers' of color experiences with the diagnostic process of autism spectrum disorder. Autism. 2023 May;27(4):876-889. doi: 10.1177/13623613221128171. Epub 2022 Nov 2. PMID 36321366
- [Background] Magana S, Parish SL, Son E. Have Racial and Ethnic Disparities in the Quality of Health Care Relationships Changed for Children With Developmental Disabilities and ASD? Am J Intellect Dev Disabil. 2015 Nov;120(6):504-13. doi: 10.1352/1944-7558-120.6.504. PMID 26505871